CLINICAL TRIAL: NCT05523791
Title: Can we Add Whey Protein Supplementation in Patients With Parkinson's Disease Without Interfering With Levodopa Response?
Brief Title: Whey Protein Supplementation in Patients With Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ospedale Generale Di Zona Moriggia-Pelascini (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4803
Record Dates: First submitted 2022-08-17; First posted 2022-08-31 (Actual); Last update posted 2022-08-31 (Actual); Status verified 2022-08

CONDITIONS: Parkinson Disease
Keywords: levodopa; whey protein supplementation; aerobic rehabilitation
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WPS (Experimental): Patients continued their standard therapy, received a standard protein redistribution dietary regimen plus a whey protein-based oral formula twice a day
  Interventions: Dietary Supplement: Fortiral
- Mg (Active Comparator): Patients continued their standard therapy, received a standard protein redistribution dietary regimen plus 2.250g of magnesium pidolate twice a day
  Interventions: Dietary Supplement: Mg++

INTERVENTIONS:
Dietary Supplement: Fortiral — Twice a day, patients took 10 g of powder containing 92.5% whey protein with 2.7% cysteine; emulsifier: soy lecithin, lactose free to be reconstituted with 150-200 ml of water.
  Arms: WPS
Dietary Supplement: Mg++ — Twice a day, patients took 2.250g of magnesium pidolate (=184 mg of Magnesium++ ione) powder twice a day to be reconstituted with 150-200 ml of water
  Arms: Mg

SUMMARY:
Many dietary supplementations are available to help people in balancing the protein intake and overcoming muscle mass loss. However, most of the products contain protein and could potentially affect levodopa action in people with Parkinson's disease (PWPD). The study aims at verify if whey protein supplementation interferes with dopamine replacement therapy efficacy in PWPD admitted at the clinic for a four weeks intensive multidisciplinary rehabilitation training.

DETAILED DESCRIPTION:
Authors performed a randomised single blind monocentric study on PWPD admitted in the rehabilitative unit of the Moriggia Pelascini Hospital for a 4-week multidisciplinary intensive aerobic rehabilitation treatment. All patients received a standard protein redistribution dietary regimen plus a whey protein-based oral formula (N=26) or Magnesium (N=25) twice daily for 28 days.

Neurological assessment and physical evaluation were conducted before (T0) and after (T1) rehabilitative treatment; dopamine replacement therapy was recorded T0 and T1 as well. The delta of changes within groups in neurological (UPDRS III) and physical (TUG, 6MW) evaluation scales was compared between groups.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of Parkinson's disease (UKBB criteria Hughes et al., 1992),
* H&Y stage 2 or 3
* presence of motor fluctuations (by means of UPDRS III item 4.3≥1)

Exclusion Criteria:

* cognitive decline

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Assessment of maintained efficacy of dopaminergic therapy in WPS group | 4 weeks
  Comparison of the deltas (T1-T0) of motor improvement (measured by UPDRS III; TUG, 6MWT) and of therapy (levodopa and LED) between the two groups.
  Eventual impact of whey protein supplementation intake would lead to lower improvement in motor scales and/or need higher dopaminergic replacement therapy doses,

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale Generale di Zona Moriggia Pelascini, Gravedona, Como, Italy

IPD SHARING:
Plan to Share IPD: Undecided